CLINICAL TRIAL: NCT02375490
Title: A Multilevel Intervention to Increase Physical Activity and Improve Healthy Eating Among Young Children (Ages 3-5) Attending Early Childcare Centres: the Healthy Start Study
Brief Title: Healthy Start to Increase Physical Activity and Improve Healthy Eating in Early Childcare Centres
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Mathieu Bélanger, Associate professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6282-15-2010/3381056-RSFS
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Pediatric Obesity
Keywords: Exercise; Eating Behavior; Preschool Child; Early Childcare Center; Obesity; Physical Literacy
MeSH Terms: conditions — Pediatric Obesity; Motor Activity; Feeding Behavior; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention arm (Experimental): The intervention arm will participate in Healthy Start.
  Interventions: Behavioral: Healthy Start
- Control arm (No Intervention): Control arm will pursue daily activities at early childcare center as usual.

INTERVENTIONS:
Behavioral: Healthy Start — Healthy Start was designed to promote physical activity and healthy eating among 3-5 year old children. Specifically, Healthy Start attempts to influence factors at the intrapersonal, interpersonal, organizational, community and physical environment and political levels. These levels of influence are targeted such that from an operational stand point, Healthy Start is composed of six interlinked components: 1) intersectoral partnerships that leads to promoting healthy weights in communities and ECC; 2) The Healthy Start guide for educators; 3) customized training, role modelling and monitoring; 4) an evidence-based resource for both families and educators; 5) supplementary resources from governmental partners; and 6) a knowledge development and exchange, and communication strategy.
  Arms: Intervention arm

SUMMARY:
Childhood obesity is one of the greatest challenges facing public health and recent evidence shows it begins in preschool aged children. It has been suggested that interventions be carried out to improve physical activity and healthy eating behaviour among young children. This study aims to fully evaluate Healthy Start, a multilevel physical activity and healthy eating intervention for preschool aged children. It is hypothesized that the Healthy Start intervention will improve both eating and physical activity behaviors of children attending early childcare centers because of its influence on multiple factors.

DETAILED DESCRIPTION:
Childhood obesity is one of the greatest challenges facing public health in the 21st century. In 2010, an estimated 43 million preschool aged children suffered from overweight or obesity and another 92 million were at risk of being overweight. From 1990 to 2010, the prevalence of overweight and obesity in children under the age of 5 increased from 4.2% to 6.7%, and it is estimated that 60 million children will suffer from being overweight by 2020. In Canada, the prevalence of obesity in preschool aged children is three times higher than the global average. Being overweight in childhood has been associated with compromised emotional health and social wellbeing. Much of the excess weight in obese children is gained before the age of 5 years and many studies indicate that adiposity tracks into childhood. Further, children who become obese before the age of 6 are at least four times more at risk of obesity in adulthood.

The problem of obesity is multifactorial, but is primarily influenced by energy intake and energy expenditure. Eating habits are established early in childhood and can be sustained for many years. Data show that only 29% of Canadian preschool aged children meet recommendations for fruit and vegetable intake and 23% for grain products. Further, 79% of 4-5 year olds consume food of little nutritional value (ex: chips, french fries, candy, chocolate, soft drinks, cake and cookies) at least once a week and other studies have demonstrated that empty calories are making up as much as 40% of their total caloric intake. Similarly, a recent review demonstrated that physical activity (PA) levels in early childcare centers (ECC) are generally low, and that time spent in sedentary state is elevated. It was estimated that children in ECC accumulate an average of 7 to 13 minutes of moderate-to-vigorous PA (MVPA) during the course of a 7 hour day. Correspondingly, recent data suggest that the prevalence of children with poor physical literacy is high and that low physical literacy competence is negatively associated with PA, cardiorespiratory fitness and weight status. These data are troubling given that sedentary and physical activity levels track over time.

Several organizations have recognized the need to counter pediatric obesity and to develop physical activity and nutrition-based interventions for pre-school populations. More than half of young Canadians between the ages of 6 months and 5 years spend around 29 hours a week in ECC, making them rich environments for implementing strategies to help children adopt healthy lifestyles. For example, one pilot study demonstrated an increase in fruit and vegetable intake following nutrition education and increased availability of healthy foods in ECC. Another intervention study integrating physical activity in all aspects of the preschool curriculum reported a 2 minute increase in classroom MVPA as assessed by accelerometer. However, both a systematic review on obesity prevention interventions in children under 5 years and another on obesity prevention policies, practice and interventions in ECC reported limited success of current interventions in positively influencing physical activity levels, dietary behaviour, or body composition. The authors suggest that the least successful interventions were unidimensional, while the most successful interventions were those with a positive impact on knowledge, abilities and competence, suggesting that interventions should be conceived based on comprehensive behaviour change models. It was also found that few interventions focused on physical activity and eating behaviour in combination, and that future interventions should target both behaviours simultaneously.

Interventions promoting healthy weight in children should encompass a broad spectrum of concerted actions and be based on best available knowledge from research and practice. Healthy Start, an intersectional multilevel physical activity and healthy eating promotion in preschool aged children, was developed on these bases. The aim of the current study is to lead a comprehensive evaluation of the Healthy Start intervention using an experimental research design.

The Intervention The population health approach is based on the concept that in order to positively influence population-level health outcomes, one needs to account for the wide range of health determinants [39], recognise the importance and complexity of potential interplay among these determinants, and reduce social and material inequities. Further, interventions adhering to principles of the population health approach rely on best evidence available, stimulate intersectoral collaborations, and provide opportunities for all potential stakeholders to be meaningfully engaged in its development. Several models based on the population health approach have been developed to help guide interventions. These models provide holistic conceptual frameworks which, similar to ecological models, suggest that interventions include a series of concerted actions capable of targeting all levels of influence, including the intrapersonal (biological and psychological), interpersonal (social and cultural), organizational, community, physical environment and political levels.

The conceptual development of Healthy Start is based on this population health approach; it includes strategies to guide each level of influence with the aim of improving children physical activity and dietary behaviours. The development of Healthy Start was a concerted action including academicians, community groups, educators, parents, and government representatives. Their effort, supported by Phase I of federal funding from the Public Health Agency of Canada (2007-2010), also involved pilot testing and improving the intervention which was designed to be multilevel, inclusive, intersectoral. It is also noteworthy, that Healthy Start was developed to be linguistically and culturally adapted to cater to both official linguistic groups in Canada, which is important since it has been documented that to be effective, it is not sufficient for interventions to be translated, they must also have been adapted for the target population.

Therefore, Healthy Start was designed to promote physical activity and healthy eating among Anglophone and Francophone 3-5 year old children in ECC (i.e. licenced daycares, preschools and pre-kindergarten programs). The vision of Healthy Start is to ensure young children eat healthily and are physically active every day. The mission is to encourage and enable families and educators to integrate physical activity and healthy eating in the daily lives of young children. Specifically, Healthy Start attempts to influence factors at the intrapersonal (ex: eating and physical activity behaviour of children), interpersonal (ex: educators and parents), organizational (ex. child care centres), community (ex: community organization involvement), and physical environment and political levels (ex: built environment and policies). These levels of influence are targeted such that from an operational stand point, Healthy Start is composed of six interlinked components (more details presented in Figure 1) : 1) intersectoral partnerships conducive to participatory action that leads to promoting healthy weights in communities and ECC; 2) The Healthy Start guide for educators on implementing healthy eating and physical activity in young children; 3) customized training, role modelling and monitoring of Healthy Start in early learning centres; 4) an evidence-based resource, LEAP-GRANDIR which contains material for both families and educators; 5) supplementary resources from governmental partners; and 6) a knowledge development and exchange (KDE), and communication strategy involving social media and web-resources to raise awareness and mobilize grassroots organizations and communities.

Study Objectives

It is hypothesized that, in comparison to usual practice, exposure to the Healthy Start intervention will lead to improved opportunities for physical activities and healthy eating and to increased physical activity and healthier eating among children. The specific study objectives are to:

1. Investigate whether the Healthy Start intervention leads to increases in child care centre-provided opportunities for physical activity and healthy eating;
2. Investigate whether the Healthy Start intervention leads to increases in physical activity levels and healthy eating behaviours among children; and
3. Investigate whether the Healthy Start intervention leads to improvements in physical literacy among children.

ELIGIBILITY:
Inclusion Criteria:

* Early childcare center must prepare and provide meals for lunch

Exclusion Criteria:

* Any early childcare center that has already received a physical activity or nutrition promoting intervention in the past to avoid underestimating the effect of the Healthy Start intervention
* For feasibility reasons, the number of children attending the early childcare center also serves as an exclusion criterion; centers with less than 20 children from the ages of 3 to 5 are not considered

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 897 (Actual)
Dates: Start 2013-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Physical Activity Level | The intervention spans a period of 6 months. Outcomes are measured before and after intervention.
  Children's physical activity levels are obtained using an Actical accelerometer worn during attendance of ECC for five consecutive days. Accelerometers represent an objective and valid method of measuring physical activity in preschool aged children.
Physical Literacy | The intervention spans a period of 6 months. Outcomes are measured before and after intervention.
  Physical literacy and gross motor skills of children will be measured using the Test of Gross Motor Development (TGMD-II). The TGMD-II is a standardized test designed to assess the gross motor functioning in children aged 3 through 10 years
Dietary Intake | The intervention spans a period of 6 months. Outcomes are measured before and after intervention.
  Intake analysis provides information on the intake of calories, macronutrients and micronutrients in children attending the centers. This method has been extensively used in studies concerning school-aged children and is considered the most precise measurement of dietary intake. In this study, intake analysis is done using the photography-assisted weighted plate waste method centers.

SECONDARY OUTCOMES:
Early Childcare Center Practices and Policies for Physical Activity and Nutrition | The intervention spans a period of 6 months. Outcomes are measured before and after intervention.
  Dietary and physical activity practices and policies in ECC are measured using the Nutrition and Physical Activity Self-Assessment of Child Care (NAP SACC), filled out independently by two research assistants in each ECC.

OTHER OUTCOMES:
Body Mass Index | The intervention spans a period of 6 months. Outcomes are measured before and after intervention.
  Height and weight are measured using a standardized protocol. A composite outcome measure, body mass index (BMI), is calculated using the ratio of weight (kg) and squared height (m2) and will be used to determine if children are overweight or obese by following the International Obesity Task Force thresholds as recommended.
Waist circumference | The intervention spans a period of 6 months. Outcomes are measured before and after intervention.
  Waist circumference is measured using a standardized protocol. Two measures of waist circumference to the nearest 0.1cm are obtain for each participant. If discrepancies greater than 0.5 cm are observed between the two measures, a third measure is obtained. The average of the two closest measures is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Leis, PhD, Principal Investigator — University of Saskatchewan; Mathieu Bélanger, PhD, Principal Investigator — Université de Sherbrooke; Louise Humbert, PhD, Principal Investigator — University of Saskatchewan; Hassan Vatanparast, PhD, Principal Investigator — University of Saskatchewan; Nazeem Muhajarine, PhD, Principal Investigator — University of Saskatchewan
Locations (2):
- Canada (2):
  - Centre de formation médicale du Nouveau-Brunswick, Moncton, New Brunswick
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Onis M, Blossner M, Borghi E. Global prevalence and trends of overweight and obesity among preschool children. Am J Clin Nutr. 2010 Nov;92(5):1257-64. doi: 10.3945/ajcn.2010.29786. Epub 2010 Sep 22. PMID 20861173
- [Background] Shields M. Overweight and obesity among children and youth. Health Rep. 2006 Aug;17(3):27-42. PMID 16981484
- [Background] Reilly JJ, Methven E, McDowell ZC, Hacking B, Alexander D, Stewart L, Kelnar CJ. Health consequences of obesity. Arch Dis Child. 2003 Sep;88(9):748-52. doi: 10.1136/adc.88.9.748. PMID 12937090
- [Background] Gardner DS, Hosking J, Metcalf BS, Jeffery AN, Voss LD, Wilkin TJ. Contribution of early weight gain to childhood overweight and metabolic health: a longitudinal study (EarlyBird 36). Pediatrics. 2009 Jan;123(1):e67-73. doi: 10.1542/peds.2008-1292. PMID 19117849
- [Background] Nader PR, O'Brien M, Houts R, Bradley R, Belsky J, Crosnoe R, Friedman S, Mei Z, Susman EJ; National Institute of Child Health and Human Development Early Child Care Research Network. Identifying risk for obesity in early childhood. Pediatrics. 2006 Sep;118(3):e594-601. doi: 10.1542/peds.2005-2801. PMID 16950951
- [Background] Quattrin T, Liu E, Shaw N, Shine B, Chiang E. Obese children who are referred to the pediatric endocrinologist: characteristics and outcome. Pediatrics. 2005 Feb;115(2):348-51. doi: 10.1542/peds.2004-1452. PMID 15687443
- [Background] Guo SS, Huang C, Maynard LM, Demerath E, Towne B, Chumlea WC, Siervogel RM. Body mass index during childhood, adolescence and young adulthood in relation to adult overweight and adiposity: the Fels Longitudinal Study. Int J Obes Relat Metab Disord. 2000 Dec;24(12):1628-35. doi: 10.1038/sj.ijo.0801461. PMID 11126216
- [Background] Freedman DS, Khan LK, Serdula MK, Dietz WH, Srinivasan SR, Berenson GS. The relation of childhood BMI to adult adiposity: the Bogalusa Heart Study. Pediatrics. 2005 Jan;115(1):22-7. doi: 10.1542/peds.2004-0220. PMID 15629977
- [Background] Hill JO, Melanson EL. Overview of the determinants of overweight and obesity: current evidence and research issues. Med Sci Sports Exerc. 1999 Nov;31(11 Suppl):S515-21. doi: 10.1097/00005768-199911001-00005. PMID 10593521
- [Background] Birch LL, Fisher JO. Development of eating behaviors among children and adolescents. Pediatrics. 1998 Mar;101(3 Pt 2):539-49. PMID 12224660
- [Background] Pabayo R, Spence JC, Casey L, Storey K. Food consumption patterns in preschool children. Can J Diet Pract Res. 2012 Summer;73(2):66-71. doi: 10.3148/73.2.2012.66. PMID 22668839
- [Background] Reedy J, Krebs-Smith SM. Dietary sources of energy, solid fats, and added sugars among children and adolescents in the United States. J Am Diet Assoc. 2010 Oct;110(10):1477-84. doi: 10.1016/j.jada.2010.07.010. PMID 20869486
- [Background] Langlois K, Garriguet D. Sugar consumption among Canadians of all ages. Health Rep. 2011 Sep;22(3):23-7. PMID 22106786
- [Background] Reilly JJ, Kelly J. Long-term impact of overweight and obesity in childhood and adolescence on morbidity and premature mortality in adulthood: systematic review. Int J Obes (Lond). 2011 Jul;35(7):891-8. doi: 10.1038/ijo.2010.222. Epub 2010 Oct 26. PMID 20975725
- [Background] Temple VA, Naylor PJ, Rhodes RE, Higgins JW. Physical activity of children in family child care. Appl Physiol Nutr Metab. 2009 Aug;34(4):794-8. doi: 10.1139/H09-061. PMID 19767816
- [Background] Hardy LL, Reinten-Reynolds T, Espinel P, Zask A, Okely AD. Prevalence and correlates of low fundamental movement skill competency in children. Pediatrics. 2012 Aug;130(2):e390-8. doi: 10.1542/peds.2012-0345. Epub 2012 Jul 23. PMID 22826575
- [Background] Gentier I, D'Hondt E, Shultz S, Deforche B, Augustijn M, Hoorne S, Verlaecke K, De Bourdeaudhuij I, Lenoir M. Fine and gross motor skills differ between healthy-weight and obese children. Res Dev Disabil. 2013 Nov;34(11):4043-51. doi: 10.1016/j.ridd.2013.08.040. Epub 2013 Sep 13. PMID 24036485
- [Background] Fisher A, Reilly JJ, Kelly LA, Montgomery C, Williamson A, Paton JY, Grant S. Fundamental movement skills and habitual physical activity in young children. Med Sci Sports Exerc. 2005 Apr;37(4):684-8. doi: 10.1249/01.mss.0000159138.48107.7d. PMID 15809570
- [Background] Lubans DR, Morgan PJ, Cliff DP, Barnett LM, Okely AD. Fundamental movement skills in children and adolescents: review of associated health benefits. Sports Med. 2010 Dec 1;40(12):1019-35. doi: 10.2165/11536850-000000000-00000. PMID 21058749
- [Background] Williams HG, Pfeiffer KA, O'Neill JR, Dowda M, McIver KL, Brown WH, Pate RR. Motor skill performance and physical activity in preschool children. Obesity (Silver Spring). 2008 Jun;16(6):1421-6. doi: 10.1038/oby.2008.214. Epub 2008 Apr 3. PMID 18388895
- [Background] Kjonniksen L, Torsheim T, Wold B. Tracking of leisure-time physical activity during adolescence and young adulthood: a 10-year longitudinal study. Int J Behav Nutr Phys Act. 2008 Dec 29;5:69. doi: 10.1186/1479-5868-5-69. PMID 19113990
- [Background] Telama R, Yang X, Viikari J, Valimaki I, Wanne O, Raitakari O. Physical activity from childhood to adulthood: a 21-year tracking study. Am J Prev Med. 2005 Apr;28(3):267-73. doi: 10.1016/j.amepre.2004.12.003. PMID 15766614
- [Background] Tammelin T. A review of longitudinal studies on youth predictors of adulthood physical activity. Int J Adolesc Med Health. 2005 Jan-Mar;17(1):3-12. doi: 10.1515/ijamh.2005.17.1.3. PMID 15900807
- [Background] Telama R. Tracking of physical activity from childhood to adulthood: a review. Obes Facts. 2009;2(3):187-95. doi: 10.1159/000222244. Epub 2009 Jun 12. PMID 20054224
- [Background] Hallal PC, Victora CG, Azevedo MR, Wells JC. Adolescent physical activity and health: a systematic review. Sports Med. 2006;36(12):1019-30. doi: 10.2165/00007256-200636120-00003. PMID 17123326
- [Background] Baur LA. Tackling the epidemic of childhood obesity. CMAJ. 2009 Mar 31;180(7):701-2. doi: 10.1503/cmaj.090196. No abstract available. PMID 19332745
- [Background] Larson N, Ward DS, Neelon SB, Story M. What role can child-care settings play in obesity prevention? A review of the evidence and call for research efforts. J Am Diet Assoc. 2011 Sep;111(9):1343-62. doi: 10.1016/j.jada.2011.06.007. PMID 21872698
- [Background] Story M, Kaphingst KM, French S. The role of child care settings in obesity prevention. Future Child. 2006 Spring;16(1):143-68. doi: 10.1353/foc.2006.0010. PMID 16532662
- [Background] Trost SG, Fees B, Dzewaltowski D. Feasibility and efficacy of a "move and learn" physical activity curriculum in preschool children. J Phys Act Health. 2008 Jan;5(1):88-103. doi: 10.1123/jpah.5.1.88. PMID 18209256
- [Background] Hesketh KD, Campbell KJ. Interventions to prevent obesity in 0-5 year olds: an updated systematic review of the literature. Obesity (Silver Spring). 2010 Feb;18 Suppl 1:S27-35. doi: 10.1038/oby.2009.429. PMID 20107458
- [Background] Evans RG, Barer ML, Hertzman C, Roos NP, Wolfson M. Why are some books important (and others not)? Can J Public Health. 2010 Nov-Dec;101(6):433-5. doi: 10.1007/BF03403957. PMID 21370774
- [Background] Kumanyika S, Jeffery RW, Morabia A, Ritenbaugh C, Antipatis VJ; Public Health Approaches to the Prevention of Obesity (PHAPO) Working Group of the International Obesity Task Force (IOTF). Obesity prevention: the case for action. Int J Obes Relat Metab Disord. 2002 Mar;26(3):425-36. doi: 10.1038/sj.ijo.0801938. No abstract available. PMID 11896500
- [Background] Huynen MM, Martens P, Hilderink HB. The health impacts of globalization: a conceptual framework. Global Health. 2005 Aug 3;1:14. doi: 10.1186/1744-8603-1-14. PMID 16078989
- [Background] Kao HF, Hsu MT, Clark L. Conceptualizing and critiquing culture in health research. J Transcult Nurs. 2004 Oct;15(4):269-77. doi: 10.1177/1043659604268963. PMID 15359059
- [Background] Adolph AL, Puyau MR, Vohra FA, Nicklas TA, Zakeri IF, Butte NF. Validation of uniaxial and triaxial accelerometers for the assessment of physical activity in preschool children. J Phys Act Health. 2012 Sep;9(7):944-53. doi: 10.1123/jpah.9.7.944. Epub 2011 Dec 27. PMID 22207582
- [Background] Pate RR, O'Neill JR, Mitchell J. Measurement of physical activity in preschool children. Med Sci Sports Exerc. 2010 Mar;42(3):508-12. doi: 10.1249/MSS.0b013e3181cea116. PMID 20068498
- [Background] Pfeiffer KA, McIver KL, Dowda M, Almeida MJ, Pate RR. Validation and calibration of the Actical accelerometer in preschool children. Med Sci Sports Exerc. 2006 Jan;38(1):152-7. doi: 10.1249/01.mss.0000183219.44127.e7. PMID 16394968
- [Background] Esliger DW, Tremblay MS. Technical reliability assessment of three accelerometer models in a mechanical setup. Med Sci Sports Exerc. 2006 Dec;38(12):2173-81. doi: 10.1249/01.mss.0000239394.55461.08. PMID 17146326
- [Background] Colley R, Connor Gorber S, Tremblay MS. Quality control and data reduction procedures for accelerometry-derived measures of physical activity. Health Rep. 2010 Mar;21(1):63-9. PMID 20426228
- [Background] Colley RC, Garriguet D, Janssen I, Craig CL, Clarke J, Tremblay MS. Physical activity of Canadian children and youth: accelerometer results from the 2007 to 2009 Canadian Health Measures Survey. Health Rep. 2011 Mar;22(1):15-23. PMID 21510586
- [Background] Crouter SE, Schneider PL, Karabulut M, Bassett DR Jr. Validity of 10 electronic pedometers for measuring steps, distance, and energy cost. Med Sci Sports Exerc. 2003 Aug;35(8):1455-60. doi: 10.1249/01.MSS.0000078932.61440.A2. PMID 12900704
- [Background] Schneider PL, Crouter SE, Lukajic O, Bassett DR Jr. Accuracy and reliability of 10 pedometers for measuring steps over a 400-m walk. Med Sci Sports Exerc. 2003 Oct;35(10):1779-84. doi: 10.1249/01.MSS.0000089342.96098.C4. PMID 14523320
- [Background] Schneider PL, Crouter S, Bassett DR. Pedometer measures of free-living physical activity: comparison of 13 models. Med Sci Sports Exerc. 2004 Feb;36(2):331-5. doi: 10.1249/01.MSS.0000113486.60548.E9. PMID 14767259
- [Background] Blakeway SF, Knickrehm ME. Nutrition education in the Little Rock school lunch program. J Am Diet Assoc. 1978 Apr;72(4):389-91. PMID 565371
- [Background] Lee HS, Lee KE, Shanklin CW. Elementary students' food consumption at lunch does not meet recommended dietary allowance for energy, iron, and vitamin A. J Am Diet Assoc. 2001 Sep;101(9):1060-3. doi: 10.1016/S0002-8223(01)00261-9. No abstract available. PMID 11573762
- [Background] Whatley JE, Donnelly JE, Jacobsen DJ, Hill JO, Carlson MK. Energy and macronutrient consumption of elementary school children served modified lower fat and sodium lunches or standard higher fat and sodium lunches. J Am Coll Nutr. 1996 Dec;15(6):602-7. doi: 10.1080/07315724.1996.10718636. PMID 8951738
- [Background] Nicklas TA, Liu Y, Stuff JE, Fisher JO, Mendoza JA, O'Neil CE. Characterizing lunch meals served and consumed by pre-school children in Head Start. Public Health Nutr. 2013 Dec;16(12):2169-77. doi: 10.1017/S1368980013001377. Epub 2013 May 24. PMID 23701867
- [Background] Williamson DA, Allen HR, Martin PD, Alfonso AJ, Gerald B, Hunt A. Comparison of digital photography to weighed and visual estimation of portion sizes. J Am Diet Assoc. 2003 Sep;103(9):1139-45. doi: 10.1016/s0002-8223(03)00974-x. PMID 12963941
- [Background] Randall Simpson JA, Keller HH, Rysdale LA, Beyers JE. Nutrition Screening Tool for Every Preschooler (NutriSTEP): validation and test-retest reliability of a parent-administered questionnaire assessing nutrition risk of preschoolers. Eur J Clin Nutr. 2008 Jun;62(6):770-80. doi: 10.1038/sj.ejcn.1602780. Epub 2007 Jun 6. PMID 17554250
- [Background] Benjamin SE, Neelon B, Ball SC, Bangdiwala SI, Ammerman AS, Ward DS. Reliability and validity of a nutrition and physical activity environmental self-assessment for child care. Int J Behav Nutr Phys Act. 2007 Jul 5;4:29. doi: 10.1186/1479-5868-4-29. PMID 17615078
- [Background] Benjamin SE, Ammerman A, Sommers J, Dodds J, Neelon B, Ward DS. Nutrition and physical activity self-assessment for child care (NAP SACC): results from a pilot intervention. J Nutr Educ Behav. 2007 May-Jun;39(3):142-9. doi: 10.1016/j.jneb.2006.08.027. PMID 17493564
- [Background] Trost SG, Messner L, Fitzgerald K, Roths B. Nutrition and physical activity policies and practices in family child care homes. Am J Prev Med. 2009 Dec;37(6):537-40. doi: 10.1016/j.amepre.2009.09.020. PMID 19944921
- [Background] Monasta L, Lobstein T, Cole TJ, Vignerova J, Cattaneo A. Defining overweight and obesity in pre-school children: IOTF reference or WHO standard? Obes Rev. 2011 Apr;12(4):295-300. doi: 10.1111/j.1467-789X.2010.00748.x. PMID 20492539
- [Derived] Abobakar L, Engler-Stringer R, Leis A, Vatanparast H. Evaluation of the impact of the Healthy Start/Depart Sante intervention on improving menu planning practices and improving the congruence between planned menus and actual food served in Saskatchewan childcare centres. Prev Med Rep. 2021 May 25;23:101403. doi: 10.1016/j.pmedr.2021.101403. eCollection 2021 Sep. PMID 34136337
- [Derived] Ward S, Belanger M, Leis A. Comparison between the Healthy Start-Depart Sante online and in-person training of childcare educators to improve healthy eating and physical activity practices and knowledge of physical activity and fundamental movement skills: A controlled trial. Prev Med Rep. 2020 Nov 28;20:101264. doi: 10.1016/j.pmedr.2020.101264. eCollection 2020 Dec. PMID 33354492
- [Derived] Leis A, Ward S, Vatanparast H, Humbert ML, Chow AF, Muhajarine N, Engler-Stringer R, Belanger M. Effectiveness of the Healthy Start-Depart Sante approach on physical activity, healthy eating and fundamental movement skills of preschoolers attending childcare centres: a randomized controlled trial. BMC Public Health. 2020 Apr 19;20(1):523. doi: 10.1186/s12889-020-08621-9. PMID 32306943
- [Derived] Belanger M, Humbert L, Vatanparast H, Ward S, Muhajarine N, Chow AF, Engler-Stringer R, Donovan D, Carrier N, Leis A. A multilevel intervention to increase physical activity and improve healthy eating and physical literacy among young children (ages 3-5) attending early childcare centres: the Healthy Start-Depart Sante cluster randomised controlled trial study protocol. BMC Public Health. 2016 Apr 12;16:313. doi: 10.1186/s12889-016-2973-5. PMID 27068684